CLINICAL TRIAL: NCT05043311
Title: A Randomized, Double-blinded, Placebo-controlled Phase I/II Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of SCTV01C in Healthy Population Aged ≥18 Years Previously Vaccinated With mRNA Vaccine Against COVID-19.
Brief Title: The Safety and Immunogenicity of SCTV01C in Healthy Population Aged ≥18 Years Previously Vaccinated With mRNA COVID-19 Vaccine.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SCTV01C-01-2
Record Dates: First submitted 2021-09-12; First posted 2021-09-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled phase I/II clinical trial to evaluate the safety, tolerability and immunogenicity of SCTV01C (A Bivalent Recombinant Trimeric S Protein Vaccine against SARS-CoV-2 Variants) in healthy population aged ≥18 years previously vaccinated with mRNA vaccine against COVID-19.
  In the study, participants receive 20 µg dose or placebo, 40 µg dose or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental: 20 µg dose, 18-59 years of age (phase 1/2) (Experimental)
  Interventions: Biological: SCTV01C
- Experimental: 20 µg dose, ≥60 years of age (phase 1/2) (Experimental)
  Interventions: Biological: SCTV01C
- Experimental: 40 µg dose, 18-59 years of age (phase 1/2) (Experimental)
  Interventions: Biological: SCTV01C
- Experimental: 40 µg dose, ≥60 years of age (phase 1/2) (Experimental)
  Interventions: Biological: SCTV01C
- Placebo Comparator: Placebo, 18-59 years of age (phase 1/2) (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo Comparator: Placebo, ≥60 years of age (phase 1/2) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SCTV01C — intramuscular injection
  Arms: Experimental: 20 µg dose, 18-59 years of age (phase 1/2); Experimental: 20 µg dose, ≥60 years of age (phase 1/2); Experimental: 40 µg dose, 18-59 years of age (phase 1/2); Experimental: 40 µg dose, ≥60 years of age (phase 1/2)
Other: Placebo — intramuscular injetion
  Arms: Placebo Comparator: Placebo, 18-59 years of age (phase 1/2); Placebo Comparator: Placebo, ≥60 years of age (phase 1/2)

SUMMARY:
The objective of this study is to evaluate the safety, tolerability and immunogenicity of SCTV01C in healthy population aged ≥18 years previously vaccinated with mRNA COVID-19 vaccine.

DETAILED DESCRIPTION:
This is a Phase I/II/III, multicenter, randomized, double-blinded trial designed to evaluate the safety, tolerability and immunogenicity of SCTV01C in healthy population aged ≥18 years previously vaccinated with mRNA COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

Phase I:

Participants are eligible to be included in the study only if the following conditions are met:

1. Male or female aged ≥18 years old when signing ICF;
2. Participants that were fully vaccinated with mRNA anti-SARS-CoV-2 vaccine, and the last dose is ≥6 months away from the vaccination of this study.
3. Participants that can sign written ICF and voluntarily participate in the trial, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. Ability to read, understand, and fill in record cards;
5. Those who are clinically judged to be healthy, the results of physical examination, vital signs and laboratory tests during the screening period are normal, or although beyond the normal reference range, they are judged by investigators to be of no clinical significance;
6. Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing age are negative on screening.

Phase II:

Participants are eligible to be included in the study only if the following conditions are met:

1. Male or female aged ≥18 years old when signing ICF;
2. Participants that were fully vaccinated with mRNA anti-SARS-CoV-2 vaccine, and the last dose is ≥6 months away from the vaccination of this study.
3. Participants that can sign written ICF and voluntarily participate in the trial, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
4. Ability to read, understand, and fill in record cards;
5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, Chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
6. Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing age are negative on screening.

Exclusion Criteria:

Phase I:

A participant who conforms to any of the following criteria should not be enrolled in the study:

1. Previous diagnosis of COVID-19;
2. High-risk populations (such as medical workers, close contacts of patients with COVID-19 infection, etc.) who are more likely to be infected with SARS-Cov-2;
3. Presence of fever within 3 days before the study vaccination;
4. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or corresponding immunosuppressants;
5. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
6. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
7. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
8. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment, or plan to use immunosuppressant therapy or immunomodulatory drugs within two years after enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed.
9. Patients on antituberculosis therapy;
10. Previously or currently suffering from clinically significant cardiovascular diseases, or clinically significant disorders related to respiratory system, liver and kidney, gastrointestinal system, endocrine system, blood and lymphatic system, metabolic and skeletal systems, or malignancies, that may affect the study assessment, or cause risks during the study vaccination, or interfere with the data interpretation as determined by the investigator;
11. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
12. Participants who received any immunoglobulin or blood products in the previous 3 months, or plan to receive similar products during the study;
13. Participants who received other investigational drugs within 1 month before the study vaccination;
14. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
15. Participants received other drug used for prevention of COVID-19 (exception for previous mRNA vaccine the participant received) ;
16. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
17. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
18. Those who are pregnant or breast-feeding;
19. Those who plan to donate ovum or sperms during the study period;
20. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
21. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
22. Those who are tested positive for hepatitis B virus (HBV), hepatitis C virus (HCV), syphilis or HIV in terms of serology.

Phase II:

A participant who conforms to any of the following criteria should not be enrolled in the study:

1. Previous diagnosis of COVID-19;
2. Presence of fever within 3 days before the study vaccination;
3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or corresponding immunosuppressants;
4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment, or plan to use immunosuppressant therapy or immunomodulatory drugs within two years after enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed.
8. Patients on antituberculosis therapy;
9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (except for skin basal cell carcinoma and carcinoma in-situ of cervix) , such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
11. Participants who received any immunoglobulin or blood products in the previous 3 months, or plan to receive similar products during the study;
12. Participants who received other investigational drugs within 1 month before the study vaccination;
13. Participants who is at the acute state of disease, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
14. Participants received other drug used for prevention of COVID-19 (exception for previous mRNA vaccine the participant received) ;
15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
17. Those who are pregnant or breast-feeding;
18. Those who plan to donate ovum or sperms during the study period;
19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
21. Those who are tested positive for HIV in terms of serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse reactions in phase 1 | Day 0 to Day 7 after the study vaccination
GMT and GMI of specific IgG total antibodies against Alpha (B.1.1.7), Beta (B.1.351), Gamma (P.1) and Delta (B.1.617.2) variants of SARS-CoV-2 in phase 2 | Day 14 after the study vaccination
GMT and GMI of neutralizing antibodies titers in phase 2 | Day 14 after the study vaccination
Incidence and severity of solicited AEs in phase 2 | Day 0 to Day 7 after the study vaccination

SECONDARY OUTCOMES:
Incidence and severity of solicited adverse events in phase 1 | Day 0 to Day 7 after the study vaccination
Incidence and severity of all unsolicited adverse events in phase 1 | Day 0 to Day 28 after the study vaccination
Incidence and severity of laboratory abnormalities related adverse events in phase 1 | Day 3 after the study vaccination
Incidence and severity of serious adverse events (SAEs), adverse events of special interest (AESIs) and medically attended adverse events (MAAEs) in phase 1 | Within 180 days after the study vaccination
GMT and GMI of specific IgG total antibodies against Alpha (B.1.1.7), Beta (B.1.351), Gamma (P.1) and Delta (B 1.617.2) variants of SARS-CoV-2 in phase 1 | Day 14 after the study vaccination
GMT and GMI of neutralizing antibodies titers for Delta (B.1.617.2) variant of SARS-CoV-2 in phase 1 | Day 14 after the study vaccination
GMT and GMI of specific total IgG antibodies against Alpha (B.1.1.7), Beta (B.1.351), Gamma (P.1) and Delta (B.1.617.2) variants of SARS-CoV-2 in phase 2 | Day 180 after the study vaccinatio
GMT and GMI of neutralizing antibodies titers for Delta (B.1.617.2) variant of SARS-CoV-2 in phase 2 | Day 180 after the study vaccination
Incidence and severity of unsolicited adverse events in phase 2 | Day 0 to Day 28 after the study vaccination
Incidence and severity of SAEs, AESIs and MAAEs in phase 2 | Within 180 days after the study vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Yang Wang, Ph.D., Study Director — Sinocelltech Ltd.
Locations (1):
- Al Kuwait Hospital (Al Baraha Hospital), Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannawi S, Saifeldin L, Abuquta A, Alamadi A, Mahmoud SA, Hassan A, Liu D, Yan L, Xie L. Safety and immunogenicity of a bivalent SARS-CoV-2 protein booster vaccine, SCTV01C, in adults previously vaccinated with mRNA vaccine: a randomized, double-blind, placebo-controlled phase 1/2 clinical trial. EBioMedicine. 2023 Jan;87:104386. doi: 10.1016/j.ebiom.2022.104386. Epub 2022 Dec 5. PMID 36470077